CLINICAL TRIAL: NCT00800423
Title: Phase 3 Study of Brimonidine Tartrate Drops Efficacy in Reducing Post Operative Corneal Edema After Cataract Surgery
Brief Title: Effect of Topical Brimonidine on Post Cataract Surgery Corneal Edema
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Robinson Anat, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5189
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Corneal Edema; Visual Acuity
Keywords: corneal edema; postoperative corneal edema; central corneal thickness; visual acuity; postoperative; brimonidine; timolol; cataract surgery
MeSH Terms: conditions — Corneal Edema | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- brimonidine (Experimental): 50 patients receiving Brimonidine Tartrate drops in the operated eye: 1 drop X2 a day for 1 month.
  they will also be administered the usual medications after cataract surgery (corticosteroids and antibiotics drops)
  Interventions: Drug: Brimonidine Tartrate 0.2%
- 2 tmolol (Active Comparator): 50 patients receiving timolol maleate 0.5% drops in the operated eye
  1 drop X2 a day for 1 month. they will also be administered the usual medications after cataract surgery (corticosteroids and antibiotics drops)
  Interventions: Drug: Timolol maleate 0.5%
- 3 (No Intervention): 50 patients will not receive any additional drug to the usual medications after cataract surgery (corticosteroids and antibiotics drops)

INTERVENTIONS:
Drug: Brimonidine Tartrate 0.2% — Brimonidine Tartrate 0.2% drops
  1 drop twice a day for 1 month in the operated eye
  Other Names: ALPHAGAN P
  Arms: brimonidine
Drug: Timolol maleate 0.5% — timolol maleate 0.5% drops
  1 drop twice a day for 1 month in the operated eye
  Other Names: TILOPTIC; V-OPTIC
  Arms: 2 tmolol

SUMMARY:
Most patients undergoing cataract surgery suffer from corneal edema after the surgery.

Brimonidine drops are a well known and safe Anti-glaucoma medication. the investigators have made several clinical observations that patients receiving Brimonidine drops had a faster resolution of their corneal edema even if they had normal intra-ocular pressure.

The investigators believe that administering topical Brimonidine to patients with significant post operative corneal edema will hasten the resolution of their corneal edema.

DETAILED DESCRIPTION:
Most patients undergoing cataract surgery suffer from corneal edema after the surgery which temporarily reduces their visual acuity until corneal edema resolves over several weeks Brimonidine drops are a well known and safe Anti-glaucoma medication, used to lower intra ocular pressure.

there have been several clinical observations that patients receiving Brimonidine drops had a faster resolution of their corneal edema even in the presence of normal intra-ocular pressure.

The investigators postulated that administering topical Brimonidine to patients with significant post operative corneal edema will hasten their recovery and visual improvement.

In order to prove that Brimonidine drops contribute to faster resolution of cornel edema and visual improvement, the study will randomly compare 50 post cataract surgery patients (group A)who will be administered Brimonidine to 2 control groups (50 people in each group):

group B will be given topical timolol drops 0.5% (another well recognized anti glaucoma medication which reduces intra-ocular pressure by different mechanism than Brimonidine.

Group C will not be given any test drug. All 3 groups will receive the regular post operative medications which include corticosteroids and antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* 1 day after uneventful cataract surgery
* corneal edema (grade 2 to 3)

Exclusion Criteria:

* glaucoma
* higher than normal intraocular pressure (>23 mm Hg)
* known sensitivity or contra indication to brimonidine
* known sensitivity or contra indication to timolol
* pre operative corneal or anterior segment disease
* intraoperative complications
* major ocular pathology other than corneal that reduced vision (retinal degeneration, optic neuropathy etc.)
* pregnant women
* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
central corneal thickness in micrometer | day 0 (day of enrollment ), day 7, day 30

SECONDARY OUTCOMES:
grading of corneal edema (1-3) | day 0 (day of enrollment), day 7, day 30

CONTACTS AND LOCATIONS:
Overall Officials: Anat Robinson, MD, Principal Investigator — Rabin medical center, Clalit health services , Israel
Locations (1):
- Rabin medical center ophthalmology deparment, Petah Tikva, Israel